CLINICAL TRIAL: NCT07101068
Title: A Randomized Clinical Trial to Assess Pain and Anxiety During Infiltration Anesthesia Using Dental Anesthesia Injector Versus Conventional Syringe in Pediatric Patients
Brief Title: Assessment of Pain and Anxiety During Infiltration Anesthesia Using Dental Anesthesia Injector Versus Conventional Syringe in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: FDSU-Rec IMO12441
Record Dates: First submitted 2025-06-15; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries; Reversible Pulpitis
Keywords: Pediatric Dentistry; Local Anesthesia; Dental Anesthesia Injector; Conventional Syringe; Pain Assessment; Vasual Analogue Scale; Corah Dental Anxiety Scale; Pulse Oximeter; Split-mouth Design; Reversible Pulpitis
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This randomized, split-mouth clinical trial uses a computerized randomization system (Sealed Envelope) to allocate the two interventions: conventional anesthesia and Dental Anesthesia Injector. For each participant, one side of the mouth will receive local anesthesia via the Dental Anesthesia Injector, while the other side will receive the conventional anesthesia method. The randomization process ensures that the assignment of anesthesia methods to the right or left side is random for each participant. Allocation concealment is maintained by a third party who is not involved in data collection and manages the allocation assignments for each new participant
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Anesthesia Injector (Experimental): Topical anesthesia lidocain for 1 minute will be applied on previously dried mucosa.
  Local anesthesia administration( artican 4% +1/100,000 With extra short needles 30G-10mm ) using Dental Anesthesia injector .
  Interventions: Device: Dental Anesthesia Injector
- Conventional syringe (Active Comparator): Topical anesthesia lidocain for 1 minute will be applied on previously dried mucosa. Local anesthesia administration( artican 4% +1/100,000 With extra short needles 30G-10mm ) using conventional syringe
  Interventions: Other: conventional syringe

INTERVENTIONS:
Device: Dental Anesthesia Injector — Topical anesthesia lidocain for 1 minute will be applied on previously dried mucosa. Local anesthesia administration( artican 4% +1/100,000 With extra short needles 30G-10mm ) using Dental Anesthesia Injector.
  Arms: Dental Anesthesia Injector
Other: conventional syringe — Topical anesthesia lidocain for 1 minute will be applied on previously dried mucosa. Local anesthesia administration( artican 4% +1/100,000 With extra short needles 30G-10mm ) using conventional syringe
  Arms: Conventional syringe

SUMMARY:
This randomized controlled trial is conducted on pediatric dental patients to compare the effectiveness of local anesthesia administered using a dental anesthesia injector device versus the traditional syringe method. The study aims to assess and compare pain and anxiety levels associated with both methods, using both subjective (self-reported) and objective measures. The goal is to identify an alternative technique that minimizes pain and anxiety in pediatric dental patients.

DETAILED DESCRIPTION:
This randomized controlled split-mouth clinical trial aims to assess pain and anxiety in pediatric dental patients during and immediately after the administration of local anesthesia using a dental anesthesia injector device compared to a conventional syringe.

The study will include healthy, cooperative children aged 6 to 8 years, each having at least one vital deeply carious maxillary primary molar with signs and symptoms of reversible pulpitis on each side of the maxilla requiring buccal infiltration anesthesia prior to pulpotomy.

Each child will receive both injection techniques on separate occasions, with random assignment of the injection method to either the right or left side (split-mouth design).

To evaluate pain and anxiety, the following tools will be used:

Pain: Visual Analogue Scale (VAS) Anxiety: Corah Dental Anxiety Scale Physiological measures: Heart rate and oxygen saturation levels, recorded using a pulse oximeter Data will be collected during and immediately after the injection. The aim is to determine whether the dental anesthesia injector provides a less painful and less anxiety-inducing experience compared to the traditional syringe method.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy patients (ASA I)
* Undergoing the first dental local anesthesia experience
* Presence of one at least vital deeply carious maxillary primary molar indicated for pulpotomy on each side of maxilla
* Score 3 or 4 of Frankl scale of child behavior

Exclusion Criteria:

* Presence of gingivitis, dental abscess, facial trauma/ injury
* Administration of analgesic 48 h before randomization
* Presence of allergy from local anesthesia

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain during injection | The pain felt by patient will be assessed by Visual analogue scale, Pulse rate and Oxygen saturation at day 1 of anesthesia injection.
  The pain felt by patient will be assessed by Visual analogue scale which is a subjective scale {rating from 0 (no pain) to 10 (worst pain ) }
  Pulse rate and oxygen saturation will be assessed also which are objective tools where the normal pulse rate is from 60 to 100 beats per minute, more than normal heart rate for the patient during injection and 1 minute after means anxiety The normal Oxygen saturation of the body is from 95% up to 100% the increase in the rating of the Oxygen saturation during the injection and 1 minute after injection means that the patient feels anxiety
Anxiety felt by the patient | the scale will be used at day 1 of anesthesia injection
  Anxiety felt by the patient during dental visit will be assessed using Corah Dental Anxiety Scale which is a subjective scale consist of brief questionnaire designed to measure anxiety related to dental visits, each question has 5 answers from a to e (a) answers give rating 1 that mean least anxiety felt and (e) answers give rating 5 that mean sever anxiety. If the total rating of the 4 questions <9 means that the patient has mild anxiety. If the total rating from 15 to 20 means that the patient has sever anxiety.

SECONDARY OUTCOMES:
Need for additional anesthesia | The assessment will be done during dental visit at day 1 of anesthesia injection
  Need for additional anesthesia will be assessed by the operator if the patient feels pain and we have to administer additional anesthesia with the same concentration and the same tool of injection for the second time to treat the same tooth at same dental visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mohamed Shafik, Associate Professor, Study Director — Pediatric Dentistry department, Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Cairo Governorate
  - Faculty of dentistry, Ain Shams University, Cairo, Cairo Governorate

IPD SHARING:
Plan to Share IPD: No
Faculty of Dentistry Ain Shams university Research Ethics Committee, state that data will not be shared to preserve the confidentiality.

REFERENCES:
- [Background] Vitale MC, Gallo S, Pascadopoli M, Alcozer R, Ciuffreda C, Scribante A. Local anesthesia with SleeperOne S4 computerized device vs traditional syringe and perceived pain in pediatric patients: a randomized clinical trial. J Clin Pediatr Dent. 2023 Jan;47(1):82-90. doi: 10.22514/jocpd.2023.002. Epub 2023 Jan 3. PMID 36627224